CLINICAL TRIAL: NCT02664064
Title: Evaluation of an Online Diabetes Prevention Program Adapted for Safety Net Users
Brief Title: Evaluation of Prevent in Underserved Populations
Acronym: PUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omada Health, Inc. (Industry)
Collaborators: Kresge Foundation (Unknown); California HealthCare Foundation (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WIRB20152184
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Prediabetes; Overweight; Obesity
Keywords: prediabetes, weight loss, behavior modification
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- online Diabetes Prevention Program (Experimental): Participants will receive access to a 12-month online diabetes prevention program modeled after the CDC DPP curriculum. Participants receive online curriculum, access to a live health coach, interactive group message forums, and connected weight and activity monitoring devices.
  Interventions: Behavioral: Prevent
- Matched Control (No Intervention): A de-identified dataset of control subjects matched on age, gender, prediabetes diagnosis, body mass index, comorbidities and socioeconomic status will be cultivated for comparison to the active intervention arm.

INTERVENTIONS:
Behavioral: Prevent — Intensive behavioral counseling for diabetes prevention and healthy lifestyle management. Recipients have access to online curriculum, a live health coach, group-based communication forums, and connected technology to track weight and physical activity.
  Arms: online Diabetes Prevention Program

SUMMARY:
The goal of this study is to evaluate an online Diabetes Prevention Program adapted for patients with prediabetes in safety net health care settings.

DETAILED DESCRIPTION:
The Diabetes Prevention Program (DPP) demonstrated that intensive behavioral counseling is a successful approach to reduce the risk of developing diabetes in patients with prediabetes. While the DPP lifestyle intervention was successful and group based adaptations of the DPP have positive results, scalable alternatives that allow for even broader reach are necessary. Omada Health has developed an online, group-based, recognized DPP program (Prevent). The goal of this study is to evaluate a literacy-adapted version of Prevent for patients with prediabetes in safety net health care settings.

ELIGIBILITY:
Inclusion Criteria:

* is receiving care at one of the three participating locations
* prediabetes diagnosis confirmed by lab tests
* age 18-75 at screening
* Not insured, Medicaid insured, or safety net health plan insured
* Comfortable speaking/reading English or Spanish at 5th grade level
* Body Mass Index greater or equal to 24
* Able to access the internet weekly by computer or smartphone
* Able to engage in physical activity of at least moderate intensity
* Able and willing to give informed consent to participate

Exclusion Criteria:

* diagnosed with Type 1 or 2 Diabetes Mellitus
* taking insulin, metformin or other hypoglycemic agent
* pregnant or planning to become pregnant during trial period
* unstable life conditions that would preclude full program participation
* acute, unstable medical or mental health conditions that would preclude program participation
* inability to engage in physical activity of at least moderate intensity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
% Weight Loss | baseline, 6 months, 12 months
  Percentage of body weight loss

SECONDARY OUTCOMES:
HbA1c | baseline, 6 months, 12 months
  fingerstick HbA1C

OTHER OUTCOMES:
Program engagement | cumulative (summary total across baseline to 12 months)
  Cumulative number of points of engagement with the online program

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Cousineau, DrPh, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - LAC+USC Medical Center, Los Angeles, California
  - Northeast Valley Health Corporation, San Fernando, California
  - Providence Medical Group-Monroe Clinic, Monroe, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Omada is a San Francisco-based healthcare technology company that is pioneering the field of digital behavioral medicine, to fulfill our mission of inspiring and enabling people everywhere to live free of chronic disease. — http://omadahealth.com